CLINICAL TRIAL: NCT03352882
Title: Impact of Transjugular Intrahepatic Portosystemic Shunts on Liver Stiffness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 826196; U54CA193417 (NIH)
Record Dates: First submitted 2017-10-04; First posted 2017-11-24 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Portal Hypertension; Liver Fibroses
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Open Label (Other): All enrolled participants will undergo hepatic ultrasound with acoustic radiation force impulse (ARFI) before and 30 days after creation of TIPS.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Hepatic ultrasound using gray scale, color Doppler, and spectral Doppler imaging to evaluate hepatic vein and portal vein patency, direction and velocity of flow respectively. ARFI will be performed in the right hepatic lobe. Three measurements of stiffness (m/s) will be performed and the mean value recorded.

SUMMARY:
Pilot study examining changes in liver stiffness measured by ultrasound before and after TIPS creation

DETAILED DESCRIPTION:
Single arm pilot study of adults ≥18yo investigating changes in liver stiffness as measured by ultrasound acoustic radiation force impulse (ARFI) before and after creation of TIPS. Duration of participation is 30 days from TIPS creation. TIPS creation with Viatorr stent graft will be in accordance with its FDA-approved indication for symptomatic portal hypertension and per the manufacturer's instructions for use. Liver stiffness will be measured on pre-TIPS and post-TIPS ultrasounds using Phillips Epiq Ultrasound systems equipped with ElastPQ ultrasound shear wave elastography. Both ultrasounds will be performed at times which are standard of care before and after TIPS creation. Primary objectives include liver stiffness as measured by ultrasound acoustic radiation force impulse (ARFI) before and after creation of TIPS. Secondary objectives include change in portosystemic gradient, clinical success as measured by difference in frequency of repeat paracentesis post-TIPS or freedom from recurrence of variceal bleeding and rate of hepatic encephalopathy. Exploratory objectives include serum biomarkers of liver stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic portal hypertension secondary to cirrhosis undergoing elective outpatient TIPS
* Age >18, Age <80
* Capable of giving informed consent

Exclusion Criteria:

* Coagulopathy defined as international normalized ration (INR) >2 which cannot be corrected with fresh frozen plasma
* Platelet count <50,000/microliter, which cannot be corrected with platelet transfusion
* BMI >35 and/or cirrhosis due to non-alcoholic steatohepatitis (due to inaccurate elastography measurements in patients with fatty liver)
* Urgent or emergent TIPS for bleeding
* Portal vein thrombosis with in the main, 1st, or 2nd order branches of the portal vein
* Hepatic vein thrombosis (ie no Budd Chiari syndrome)
* Excessive alcohol use defined as more than 2 oz in 24 hours on any individual day within the last 30 days
* Inability to provide informed consent
* Pregnant or nursing women
* Enrollment in concurrent therapeutic trial for symptomatic portal hypertension

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Forde, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 51 [51 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1
Childs-Pugh Score [Number; unit: units on a scale] — The Child-Pugh score is a system for assessing the prognosis of chronic liver disease, primarily cirrhosis. It provides a forecast of the increasing severity of liver disease and expected survival rate.The score is determined by five clinical measures of liver disease. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe. The five clinical measures are:
  * total bilirubin
  * serum albumin
  * prothrombin time, prolongation(s) or INR
  * ascites
  * hepatic encephalopathy
  The Childs-Pugh score ranges from 5 to 15 and a higher score indicates greater severity of liver disease.
  units on a scale | 8

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Liver Stiffness
Description: The primary study endpoint will be decrease in liver stiffness following TIPS creation as measured by ARFI using mean propagation velocity values in meters per second. Mean normal values and mean values indicating severe fibrosis range about 0.8-1.7 m/s and about 1-3.4 m/s respectively. We hypothesize TIPS creation will reduce the liver stiffness by > 50%. Change in liver stiffness will be correlated to change in PSG.
Time Frame: Pre-TIPS and 30 days Post-TIPS creation
Population: This study was terminated early due to low enrollment. Only 1 subject was ever enrolled and as such no data analysis was conducted.
Arm/Group | Open Label
Number analyzed (Participants) | 0

2. Secondary Outcome: PSG (mm hg) and ARFI (m/s) Correlation
Description: Baseline PSG (mm Hg) correlation to baseline liver stiffness by ultrasound ARFI (m/s)
Time Frame: Pre-TIPS and 30 days Post-TIPS creation
Population: as for outcome 1
Arm/Group | Open Label
Number analyzed (Participants) | 0

3. Secondary Outcome: Frequency of Paracentesis and Recurrence of Variceal Bleeding
Description: Difference in frequency of paracentesis and freedom from recurrence of variceal bleeding at 30 days and 12 months post-TIPS placement
Time Frame: 30 days Post-TIPS and 12 months Post-TIPS creation
Population: as for outcome 1
Arm/Group | Open Label
Number analyzed (Participants) | 0

4. Secondary Outcome: Hyaluronic Acid and ARFI Correlation
Description: Correlation of hyaluronic acid, a serum marker of liver stiffness, with baseline ARFI measurements, non-invasive radiographic assessment of liver stiffness
Time Frame: Pre-TIPS and 30 days Post-TIPS creation
Population: as for outcome 1
Arm/Group | Open Label
Number analyzed (Participants) | 0

5. Secondary Outcome: Tissue Inhibitor of Metalloproteinase-1 and ARFI Correlation
Description: Correlation of tissue inhibitor of metalloproteinase-1, a serum marker of liver stiffness, with baseline ARFI measurements, non-invasive radiographic assessment of liver stiffness
Time Frame: Pre-TIPS and 30 days Post-TIPS creation
Population: as for outcome 1
Arm/Group | Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 30 days
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03352882/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03352882/ICF_001.pdf